CLINICAL TRIAL: NCT00869024
Title: AsseSsment of Efficacy, Safety and Utility of intRa myocardiAl iNjection of Stem Cells in Patients With End Stage Heart Failure Undergoing LVAD Implantation (ASSURANCE)
Brief Title: Stem Cell Therapy in Patients With Severe Heart Failure & Undergoing Left Ventricular Assist Device Placement
Acronym: ASSURANCE
Status: Completed | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: University of Minnesota (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1106M00401
Record Dates: First submitted 2009-03-24; First posted 2009-03-25 (Estimated); Results first posted 2020-03-13 (Actual); Last update posted 2020-03-13 (Actual); Status verified 2020-02

CONDITIONS: Heart Failure
Keywords: Heart failure; Left ventricular assist device; Stem cells
MeSH Terms: conditions — Heart Failure

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Stem Cell therapy (Experimental): Intramyocardial Delivery of Bone Marrow Derived Mononuclear Cells in Patients with Severe LV Dysfunction and LVAD Support
  Interventions: Biological: Intramyocardial Delivery of Bone Marrow Derived Mononuclear Cells
- Placebo (Placebo Comparator): Intramyocardial Delivery Placebo solution into Patients with Severe LV Dysfunction and LVAD Support
  Interventions: Biological: Intramyocardial Delivery of Bone Marrow Derived Mononuclear Cells

INTERVENTIONS:
Biological: Intramyocardial Delivery of Bone Marrow Derived Mononuclear Cells — Ten separate injections will be delivered into the LV free wall (20 X 106 cells / 400 micro lit).

SUMMARY:
The purpose of this study is to determine if the delivery of cells just after implantation of left ventricular assist device will help to improve the pumping function of your heart and minimize heart enlargement in the future.

The cells will be obtained by aspiration or withdrawal of fluid from your bone marrow from your pelvic bone using a needle and syringe. This would not take place until 24-48 hours prior to your planned left ventricular assist device implantation. During the surgery the surgeons will inject the prepared cells that were taken from your bone marrow and inject it into your heart muscle.

This study will test whether receiving your own bone marrow cells directly into your heart will help your heart to recover function after placement of a left ventricular assist device.

DETAILED DESCRIPTION:
Patients who meet the inclusion and exclusion criteria and agree to participate will be enrolled in the study. All the patients will have a baseline EKG, Laboratory tests, 2D ECHO and PET/CT imaging.Day prior to the LVAD implantation all the patients will undergo bone marrow aspiration. Bone marrow aspirate will be processed according to the protocols used by that facility. After processing, the bone marrow mononuclear cells will then be suspended in 2ml of 5% human serum albumin and labeled per the standard protocol of the facility.

Patients will be randomized in a 2:1 fashion either to receive cells or 5% serum albumin. Under general anesthesia using the standard techniques the HeartMate II (LVAD) will be placed. The LVAD will be inserted into the LV apex (with removal of 2 x 2 cm ventricular core). The tissue core will be processed for RNA isolation and morphological analysis. CV surgeon will inject either the cells or placebo directly in to the myocardium in the LAD territory. Ten separate injections will be delivered into the LV free wall (20 X 106 cells / 400 micro lit). The injection sites will be marked with Titanium surgical clips. Subjects will be managed at all times by the current standard of care in this hospital for the patients with an LVAD. Routine postoperative care procedures will be followed with close follow-up for dysrrhythmias or signs of infection.

Tissue sample from the core of the left ventricular apex removed at the time of implantation of LVAD will be compared with the myocardium (marked with the surgical clips) from the explanted heart at the time of transplantation. These samples from the experimental subjects and control hearts will be examined for morphology for interstitial fibrosis, hypertrophy, myocyte diameter and myocytolysis as well as for gene expression using RT-PCR.

Research-related follow-up will take place at weeks 2, 4, 6, 8 and months 6, 12, 18 and 24 after LVAD implant at the Clinical Trial Center of the Cardiology Division at the University of Minnesota. Patients will be examined by the PI or Sub-I at each visit. Follow up data to be obtained at these clinic visits is outlined in the protocol

ELIGIBILITY:
Inclusion Criteria:

1. Severe LV dysfunction with EF < 30% with cardiomyopathy ( Ischemic and non ischemic)
2. NYHA Class III and IV
3. No revascularization options available
4. LVAD placement as destination therapy or bridging to transplantation
5. Age between 18-80 years

Exclusion Criteria:

1. History of recent malignancy( less than one year) .
2. Unstable hemodynamics at the time of the implant; defined by need for increasing vasopressor medication in the last 24 hours or blood pressure < 70 systolic, or cardiac index < 1.3 liters/min.
3. Coronary anatomy suitable for revascularization at the time of surgery
4. Pregnancy confirmed by positive urine test
5. Lactating mothers
6. Renal failure with serum creatinine >3.0, or are receiving chronic dialysis support.
7. Inability to undergo PET/CT imaging.
8. A history of any significant recent bleeding disorder or coagulation profile of concern for acute bleeding, such as INR >2.0 (not on anticoagulant), platelet count <100,000, or hemoglobin <8.0 gr/dl.
9. Patients with known infectious disease (Hepatitis, HIV) etc.
10. Patients with three times or more of the upper limits of normal enzymes.

    -

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 25 (Actual)
Dates: Start 2011-11-10 (Actual); Primary Completion 2016-03-29 (Actual); Study Completion 2016-03-29 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Ganesh Raveendran, MD, Principal Investigator — University of Minnesota
Locations (1):
- University Of Minnesota, Minneapolis, Minnesota, United States

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Stem Cell Therapy | Placebo
Started | 16 | 9 (One patient intent to treat, did not receive study product)
Completed | 14 | 4
Not Completed | 2 | 5
Not completed — Death | 2 | 3
Not completed — Lost to Follow-up | 0 | 1
Not completed — Protocol Violation | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Stem Cell Therapy | Placebo | Total
Number analyzed (Participants) | 16 | 9 | 25
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0 | 0 | 0
  Between 18 and 65 years | 8 | 4 | 12
  >=65 years | 8 | 5 | 13
Age, Continuous [Mean (Standard Deviation); unit: years] | 62.3 (8.68) | 65.1 (8.6) | 63.3 (8.58)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 3 | 0 | 3
  Male | 13 | 9 | 22
Region of Enrollment [Number; unit: participants]
  United States | 16 | 9 | 25

OUTCOME MEASURES:

1. Primary Outcome: Safety of Cell Delivery
Description: Safety as measured by the total number of adverse events per group.
Time Frame: 24 months
Measure: Number; unit: adverse events
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 16 | 4
adverse events | 1 | 0

2. Primary Outcome: Improvement in Myocardial Viability by PET/CT Scan
Description: Change in LAD segments from baseline to 10 weeks. PET scan viability is reported by segment on a scale of 0-4. A score of 0, 1, or 2 are categorized as viable/healthy heart tissue and a score of 3 or 4 are categorized as not viable/scar tissue. No change or better in viability will be reported to determine safety of cell injection. Measurement is reported as number of segment that remained the same or improved were considered "safe" for stem cell injection.
Time Frame: baseline, 10 weeks
Measure: Number; unit: safe segments
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 15 | 4
safe segments
  Anterior wall base segment | 14 | 4
  Anterior wall mid segment | 14 | 4
  Anterior lateral wall base segment | 15 | 4
  Anterior lateral wall mid segment | 15 | 4

3. Primary Outcome: Combined End Points of Death
Description: Number of participants who expired during the study.
Time Frame: 24 months
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 16 | 4
Participants | 2 | 3

4. Secondary Outcome: Number of Participants Turned Down Without Meeting LVAD Stopping Rules
Description: LVAD turn-down was completed at 10 weeks. Hemodynamic measurements were taken and reported with nominal LVAD support and then again at peak exercise. LVAD turn-down protocol was followed to ensure safety of patient while turning down their LVAD support. After each turn-down we waited 10 minutes and repeated ECHO, RHC, LVAD parameters, vital signs.
  Stopping parameters for turn down:
  1. Significant symptoms (clinician judgement, although low threshold to stop test)
  2. CVP>20 or increase by more than 10 (e.g., 5 to 16)
  3. PCWP>25 or increase by more than 10 (e.g., 11 to 22)
  4. Hypotension
  5. Increase in LVIDd by >1.5 cm
  6. Aortic valve opening minimally (less than 1 in 5 beats, e.g.)
  The number of patients that could be turn-down without meeting stopping rules and were able to exercise were reported per group.
Time Frame: 10 weeks
Measure: Count of Participants; unit: Participants
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 12 | 5
Participants | 12 | 2

5. Secondary Outcome: Change in Left Ventricular Dimensions
Description: Change in left ventricular dimensions assessed by ECHO at baseline compared to 10 weeks with LVAD turn-down to 6000 RPMs.
Time Frame: 10 weeks
Measure: Mean (Standard Deviation); unit: cm
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 14 | 6
cm
  Change from baseline to 10 weeks in LVEDD | -0.49 (1.004) | -0.57 (0.76)
  Change from baseline to 10 weeks in LVESD | -0.73 (1.07) | -0.62 (0.89)

6. Secondary Outcome: Histological Assessment
Description: Data collection was insufficient for data analysis. Samples were collected but no histological analysis performed.
Time Frame: 24 months
Population: Data collection was insufficient for data analysis. Samples were collected but no histological analysis performed.
Arm/Group | Stem Cell Therapy | Placebo
Number analyzed (Participants) | 0 | 0

ADVERSE EVENTS:
Time Frame: 24 months
Description: Adverse events are classified as serious or non-serious. A serious adverse event is any AE that is:
  fatal life-threatening requires or prolongs hospital stay results in persistent or significant disability or incapacity An important medical event
Arm/Group | Stem Cell Therapy | Placebo
All-Cause Mortality (participants affected / at risk) | 2/16 | 3/9
Serious Adverse Events (participants affected / at risk) | 13/16 | 7/9
Other Adverse Events (participants affected / at risk) | 0/16 | 0/9
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Stem Cell Therapy (N=16) | Placebo (N=9)
Fever (General disorders) | 1 (2) | 1 (1)
Transient ischemic attack (Cardiac disorders) | 0 (0) | 1 (1)
Cerebrovascular accident (Cardiac disorders) | 2 (2) | 0 (0)
Increased bleeding (Blood and lymphatic system disorders) | 7 (11) | 1 (2)
Syncope (Cardiac disorders) | 1 (1) | 0 (0)
Palpitations (Cardiac disorders) | 0 (0) | 1 (1)
Increased frequency of Atrial arrhythmias (Cardiac disorders) | 2 (2) | 1 (1)
Increased frequency of Ventricular arrhythmias (Cardiac disorders) | 3 (5) | 3 (3)
Sepsis (General disorders) | 1 (1) | 1 (1)
Endocarditis (Blood and lymphatic system disorders) | 1 (1) | 0 (0)
Any infection (Infections and infestations) | 6 (8) | 3 (3)
New Liver Failure (Hepatobiliary disorders) | 0 (0) | 2 (2)
New Renal Failure (Renal and urinary disorders) | 0 (0) | 2 (2)
Any Malignancies (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 (1) | 0 (0)
Shock (General disorders) | 1 (1) | 2 (2)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes